CLINICAL TRIAL: NCT05233852
Title: A Framework to Analyze Gender Bias in the Overuse Studies Conducting in Primary Care
Brief Title: Gender Bias in the Overuse Studies Conducting in Primary Care
Acronym: OVERGEND
Status: Active, not recruiting | Type: Observational
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, José Joaquín Mira, Professor, Universidad Miguel Hernandez de Elche
Other Study IDs: PROMETEO/2021/061
Record Dates: First submitted 2022-01-18; First posted 2022-02-10 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Severe Adverse Event
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: "Do not do" recommendation — A drug prescription or procedure included in 'do not do' recommendations

SUMMARY:
The purpose of this study is to analyze whether the differences between men and women in the frequency of adverse events due to ignoring "Do not do" recommendations in primary care setting are due to biological causes or gender bias.

DETAILED DESCRIPTION:
First, using the Delphi technique, a consensus will be reached on those "Do Not Do" recommendations that should be included in the retrospective analysis study. The selection criteria for these recommendations will be if they are considered to persist in clinical practice in primary care, their relationship with factors associated with sex and gender, and if ignoring the "Do not do" recommendation could cause a serious adverse event. Second, a retrospective cohort study will be carried out in which a random selection of medical records will be reviewed to identify the frequency of adverse events due to ignoring the "Do not do" recommendations previously selected by consensus. Investigators will review a total of 1538 medical records of patients (50% of women) who attended primary care consultation from 1st January 2022 to 31st December 2022. Data source will be the electronic record management system of the autonomous community of Valencia, named ABUCASIS. Adverse events will be identified by using an activation tool used in a previous study (SOBRINA study).

ELIGIBILITY:
Inclusion Criteria:

* Attending primary care consultation from 1 January 2017 to 31 December 2019.
* Adult

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 50% women
Study Population: Adults attending primary care consultation from 1 January 2017 to 31 December 2019.
Sampling Method: Probability Sample
Enrollment: 1538 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of severe adverse events | From date of prescription until the date of first documented severe adverse event or date of death from any cause, whichever came first, assessed up to 12 months
  Number of severe adverse events due to ignore "do not do" recommendations
Number of female patients who were recommended "do not do" | From 1st January 2022 to 31 December 2022
  Number of female patients who were recommended "do not do"
Number of male patients who were recommended "do not do" | From 1st January 2022 to 31 December 2022
  Number of male patients who were recommended "do not do"

CONTACTS AND LOCATIONS:
Locations (1):
- Miguel Hernández University, Elche, Alicante, Spain

REFERENCES:
- [Derived] Mira JJ, Carratala-Munuera C, Garcia-Torres D, Soriano C, Sanchez-Garcia A, Gil-Guillen VF, Vicente MA, Perez-Jover MV, Lopez-Pineda A. Low-value practices in primary care: a cross-sectional study comparing data between males and females in Spain. BMJ Open. 2024 Nov 24;14(11):e089006. doi: 10.1136/bmjopen-2024-089006. PMID 39581714
- [Derived] Perez-Jover V, Sanchez-Garcia A, Lopez-Pineda A, Carrillo I, Mira JJ, Carratala-Munuera C. Identification of low-value practices susceptible to gender bias in primary care setting. BMC Prim Care. 2024 Jun 8;25(1):205. doi: 10.1186/s12875-024-02456-8. PMID 38851666
- [Derived] Carrillo I, Lopez-Pineda A, Perez-Jover V, Guilabert M, Vicente MA, Fernandez C, Gil-Guillen VF, Orozco-Bletran D, Chilet-Rosell E, Luzon Oliver L, Astier-Pena MP, Tella S, Carratala-Munuera C, Mira JJ. Epidemiological study on gender bias and low-value practices in primary care: a study protocol. BMJ Open. 2023 May 9;13(5):e070311. doi: 10.1136/bmjopen-2022-070311. PMID 37160394